CLINICAL TRIAL: NCT00497640
Title: CPAP Titration Using an Artificial Neural Network: A Randomized Controlled Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to lack of interest from subjects and no funding, only 1 subject signed consent but did not participate.
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Ali El Solh, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MED4890507E
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Last update posted 2020-11-25 (Actual); Status verified 2009-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: sleep apnea, titration, CPAP, neural network
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Microcephaly, Primary Autosomal Recessive, 6

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Artificial Neural Network — Use of a predicted optimal CPAP

SUMMARY:
The purpose of the study is to determine the validity of the prediction model in reducing the rate of CPAP titration failure and in achieving a shorter time to optimal pressure

DETAILED DESCRIPTION:
In order to derive the most effective pressure, CPAP titration is performed in the sleep laboratory during which the pressure is gradually increased until apneas and hypopneas are abolished in all sleep stages and in all body positions. The technique is however time consuming and labor intensive. Furthermore, the duration of the study may not be sufficient to attain this goal because of patient's poor ability to sleep in this environment or due to difficulty in attaining an appropriate pressure. A predictive algorithm based on demographic, anthropometric, and polysomnographic data was developed to facilitate the selection of a starting pressure during the overnight titration study. Yet, the performance of this model was inconsistent when validated by other centers. One of the potential reasons for the lack of reproducibility is the complex relation of behavioral processes with nonlinear attributes. In areas of complex interactions, the artificial neural network (ANN) has been found to be a more appropriate alternative to linear, parametric statistical tools due to its inherent property of seeking information embedded in relations among variables thought to be independent.

Comparison: time to achieve optimal pressure in the conventional technique versus the intervention model

ELIGIBILITY:
Inclusion Criteria:

1. patients 18 years of age and older,
2. documented OSA by sleep study defined as AHI > 5/hr

Exclusion Criteria:

1. previously treated OSA,
2. unwilling to undergo a titration study,
3. unable or unwilling to sign an informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2008-07 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Time to achieve optimal CPAP | minutes

SECONDARY OUTCOMES:
Failure Rate of CPAP titration | percentage

CONTACTS AND LOCATIONS:
Overall Officials: Ali A El Solh, MD, MPH, Principal Investigator — Sate University of New York at Buffalo
Locations (1):
- State University of New York at Buffalo, Buffalo, New York, United States

REFERENCES:
- [Background] El Solh AA, Aldik Z, Alnabhan M, Grant B. Predicting effective continuous positive airway pressure in sleep apnea using an artificial neural network. Sleep Med. 2007 Aug;8(5):471-7. doi: 10.1016/j.sleep.2006.09.005. Epub 2007 May 18. PMID 17512788